CLINICAL TRIAL: NCT06250985
Title: New Treatment of Cardiovascular Implantable Electronic Device (CIED) Infections; Immediate Reimplantation After Removal of Infected System
Brief Title: New Treatment of Cardiac Device Infections; Immediate Reimplantation After Removal of Infected System
Acronym: POET-PPM
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Henning Bundgaard, Professor, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-23033548
Record Dates: First submitted 2024-02-01; First posted 2024-02-09 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Endocarditis, Bacterial
MeSH Terms: conditions — Endocarditis, Bacterial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Immediate reimplantation (Experimental): Reimplantation in same procedure as removal of device or shortly thereafter.
  Interventions: Other: Timing of reimplantation
- Standart care (Active Comparator): Reimplantation of device in a second procedure at a later date, after infection has been stabilized/cleared
  Interventions: Other: Timing of reimplantation

INTERVENTIONS:
Other: Timing of reimplantation — Patients will be rendomized 1:1 by computer to recieve either standart care or intervention prior to removal of infected system

SUMMARY:
The goal of this randomized clinical trials is to ascertain the safety and efficacy of immediate reimplantation of cardiac electronic implantable devices in patients with endocarditis and device-infections, compared to standard care, i.e. reimplantation at a later procedure date.

The primary outcome is the occurence of the composite primary endpoint within 6 months of randomization consisting of

* Death
* Symptomatic embolism (systemic arterial embolism or pulmonary embolism)
* Bacteremia og pocket-infection
* Removal of a CIED due to new infection

ELIGIBILITY:
Inclusion Criteria:

* Culture positive or negative infection of a CIED acording to PI
* Indication for removal of device
* Clinical indication of device removal of existing device (concurrent left-sided IE is not a contraindication).
* Indication for reimplantation of new device
* A minimum of 3 days of sufficient antibiotic treatment (intravenous or oral) has been administered and/or culture negative antibiotic regimen have been adminstered until blood culture is examined.
* stabilization criteria fulfilled i.e. I) negativ blood cultures, II) WBC < 15 mia/L or reduction of min. 25% and III) CRP <50 or min. 25% reduction.

Exclusion Criteria:

* Immunoincompetence (active chemotherapy or prednisone treatment > 20mg/day
* Device-infection within last 6 months (relaps)
* Septic shock
* Stabilization criteria not fulfilled after 10 days of suficient antibiotic treatment

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Estimated)
Dates: Start 2024-04-29 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2037-12-31 (Estimated)

PRIMARY OUTCOMES:
Composite primary outcome | within 6 months of randomization
  Composite endpoint consisting of number of participants with one or more of the following events during follow-up: death, symptomatic embolism (systemic or pulmonary), bacteremia or pocket infection with same bacterial pathogen or removal of device due to new infection.

CONTACTS AND LOCATIONS:
Overall Officials: Henning Henning, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No